CLINICAL TRIAL: NCT04266444
Title: Motivation, Neuropsychological Testing and Functional Exercise in Virtual Environment for Persons With Multiple Sclerosis or Parkinson's Disease
Brief Title: Functional Exercise in Virtual Environment for Persons With Multiple Sclerosis or Parkinson's Disease
Acronym: MEFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Rehabilitation Institute, Republic of Slovenia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URIS202001
Record Dates: First submitted 2020-02-06; First posted 2020-02-12 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Parkinson Disease; Multiple Sclerosis
Keywords: exergaming; virtual reality; neuropsychological tests; motivation
MeSH Terms: conditions — Parkinson Disease; Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Level 4 (Active Comparator): 10Cubes game in virtual reality using very small bouncing blocks
  Interventions: Device: Exergaming in virtual environment
- Level 3 (Active Comparator): 10Cubes game in virtual reality using very small non-bouncing blocks
  Interventions: Device: Exergaming in virtual environment
- Level 2 (Active Comparator): 10Cubes game in virtual reality using large bouncing blocks
  Interventions: Device: Exergaming in virtual environment
- Level 1 (Active Comparator): 10Cubes game in virtual reality using large non-bouncing blocks
  Interventions: Device: Exergaming in virtual environment

INTERVENTIONS:
Device: Exergaming in virtual environment — The 10Cubes game (by I. Cikajlo) will be used. In the game, the motion of the hand, wrist and fingers is tracked by an infra-red camera (by LeapMotion, Inc.) and hand motion is reflected in the virtual environment. The software will run on a powerful computer with a 19" display. Each group will have the game set to a different level of difficulty.

SUMMARY:
The aim of the study is to optimise the hand dexterity exercising program in virtual reality (VR) for patients with multiple sclerosis and Parkinson's disease. Little research has been published on this topic, but the preliminary results are promising. Different levels of difficulty of a VR game will be tested. The patients will be assessed using neuropsychological tests of executive functions, visuospatial abilities, mental speed, flexibility and motor speed. Functional ability, coordination and cognitive abilities will also be assessed.

DETAILED DESCRIPTION:
Each patient meeting the inclusion criteria will be randomised to one of the four groups (i.e., 10cubes game difficulty level). The patients will perform five exergaming sessions, each session lasting for 1 hour, on five consecutive working days within the period of two weeks. The 10cubes task requires that all 10 cubes are moved within 2 minutes. Each patient will perform the task 5 times in succession with 1-2 minute breaks. The patients will be assessed using the Box & Blocks Test, Frontal Assessment Battery (FAB), Delis-Kaplan Executive Function System (D-KEFS) and Judgment of Line Orientation (JLO) before the first session and after the last session. In addition, the patients will fill in the Intrinsic Motivation Inventory (IMI) after each session. Based on statistical sample size calculations, the study plan is to include 80 patients with Parkinson's disease and 12 patients with multiple sclerosis randomising them separately, so that the groups will be balanced in terms of size and diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* diagnose of Parkinson's disease or multiple sclerosis;
* Mini Mental State Examination score above 24;
* preserved upper limb function;
* for Parkinson's disease patients Hoehn and Yahr scale score between 2 and 3.

Exclusion Criteria:

* any communicable disease;
* severe vision impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Change in Box & Blocks Test from baseline | Assessment at baseline and after two weeks
  Standard clinical test to assesses unilateral gross manual dexterity; the minimum possible score is 0, the maximum is 150; higher score indicates better outcome.
Change in Frontal Assessment Battery (FAB) score from baseline | Assessment at baseline and after two weeks
  Brief neuropsychological test battery to assess executive functions; the minimum possible score is 0, the maximum is 18; higher score indicates better outcome.
Intrinsic Motivation Inventory (IMI) scores | Assessment at the end of each exergaming session; median across assessments will be taken as the outcome on each subscale
  The IMI is a multidimensional measurement instrument for assessing subjective experience of a target activity. The 22-item version that consists of four subscales will be used (scores range from 7 to 49 for one scale and from 5 to 35 for three scales); higher scores indicate better outcome.

SECONDARY OUTCOMES:
Change in Delis-Kaplan Executive Function System (D-KEFS) scores from baseline | Assessment at baseline and after two weeks
  Set of nine subtests of executive functions with complex computerised scoring; higher scores indicate better outcome.
Change in Judgment of Line Orientation (JLO) | Assessment at baseline and after two weeks
  Standardized test of visuospatial skills; the minimum possible score is 0, the maximum is 30; higher score indicates better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Imre Cikajlo, PhD, Principal Investigator — University Rehabilitation Institute, Republic of Slovenia
Locations (1):
- University Rehabilitation Institute, Republic of Slovenia, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cikajlo I, Peterlin Potisk K. Advantages of using 3D virtual reality based training in persons with Parkinson's disease: a parallel study. J Neuroeng Rehabil. 2019 Oct 17;16(1):119. doi: 10.1186/s12984-019-0601-1. PMID 31623622
- [Derived] Cikajlo I, Hukic A, Udovcic Pertot A. The size and behavior of virtual objects have influence on functional exercise and motivation of persons with multiple sclerosis: a randomized study. Sci Rep. 2022 Nov 12;12(1):19375. doi: 10.1038/s41598-022-24046-3. PMID 36371421